CLINICAL TRIAL: NCT07193667
Title: CAR-T Cell Therapy in Relapsed/Refractory Autoimmune Diseases
Brief Title: CAR-T in Subjects With Relapsed/Refractory Autoimmune Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShenZhen Cell Valley (Industry)
Collaborators: First Affiliated Hospital of China Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-757-2
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Autoimmune Diseases
Keywords: CAR-T
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- relapsed/refractory autoimmune diseases (Experimental)
  Interventions: Drug: CD19 CAR-T cells were administered to patients with relapsed/refractory autoimmune diseases

INTERVENTIONS:
Drug: CD19 CAR-T cells were administered to patients with relapsed/refractory autoimmune diseases — This is a prospective, single-center, open, single-arm, dose-escalation clinical trial to evaluate the safety and efficacy of CAR-T cell therapy in patients with relapsed/refractory autoimmune diseases. Intravenous infusion will be used, and the trial procedure will be divided as follows:
  1. Screening period (D-28 to D-6):
     After subjects voluntarily sign an informed consent form, a screening period will be conducted to determine whether subjects are eligible for the trial based on inclusion and exclusion criteria.
  2. Lymphocyte depletion pretreatment (Study D-5 to Study D-3):
     Subjects will be pre-treated with Lymphocyte depletion starting 5 days prior to CAR-T cell infusion (FC regimen)
  3. Rest and Observation (Study D-2 to Study D-1):
     Follow the study procedures and perform the relevant examinations during the rest and observation period.
  4. Cell Infusion and Primary Study Endpoint Observation Period (Study D0 to W12 post-infusion):Subjects will undergo CAR-T cell infusion at 2-da

SUMMARY:
In this study, CD19 CAR-T cells were administered to patients with relapsed/refractory autoimmune diseases. This study intends to use retroviral vector-based tandem CAR-T cells targeting CD19 to treat autoimmune disease. The CAR-T cells were provided by Shenzhen Cell Valley. A study published in the New England Journal of Medicine provides strong evidence for the therapeutic potential of CD19 CAR-T therapy in autoimmune diseases. The study enrolled 15 participants, including eight with severe SLE, three with idiopathic inflammatory myositis, and four with systemic sclerosis. The median follow-up was 15 months (4 to 29 months). Data from the clinical trial showed that all patients with SLE had a remission of DORIS, all patients with idiopathic inflammatory myositis had an ACR-EULAR major clinical response, all patients with systemic sclerosis had a decrease in the EUSTAR activity index score, and all patients discontinued immunosuppressive therapy completely. The investigators look forward to expanding the use of CAR-T cells in relapsed/refractory autoimmune diseases through this safety and efficacy clinical study and greatly enhancing the quality of life for these patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, open, single-arm, dose-escalation clinical trial to evaluate the safety and efficacy of CAR-T cell therapy in patients with relapsed/refractory autoimmune diseases. Intravenous infusion will be used, and the trial procedure will be divided as follows:

1. Screening period (D-28 to D-6):

   After subjects voluntarily sign an informed consent form, a screening period will be conducted to determine whether subjects are eligible for the trial based on inclusion and exclusion criteria.
2. Lymphocyte depletion pretreatment (Study D-5 to Study D-3):

   Subjects will be pre-treated with Lymphocyte depletion starting 5 days prior to CAR-T cell infusion (FC regimen)
3. Rest and Observation (Study D-2 to Study D-1):

   Follow the study procedures and perform the relevant examinations during the rest and observation period.
4. Cell Infusion and Primary Study Endpoint Observation Period (Study D0 to W12 post-infusion):Subjects will undergo CAR-T cell infusion at 2-day intervals (Study Day 0) after lymphocyte depletion pretreatment, and post-infusion observations and safety assessments will be performed before, during, and after the cell infusion (day of infusion, days 4, 7, 10, 14, 21, and 28 post-infusion), respectively. Evaluation of efficacy: Subjects will be evaluated for efficacy on the 14th, 28th day, 8th and 12th week after CAR-T cell infusion.
5. Follow-up period (W12 to W52 after infusion):The follow-up period is for safety and efficacy evaluation. Safety follow-up: Subjects will be followed for 52 weeks after CAR-T cell infusion. Efficacy Evaluation: Subjects will be evaluated for efficacy at weeks 24, 36, and 52 after CAR-T cell infusion. In addition, the actual frequency of effectiveness evaluations may be increased at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years (including threshold) and gender;
* positive expression of CD19 in peripheral blood B cells as determined by flow cytometry;
* the function of vital organs meets the following requirements:

  1. Bone marrow function needs to meet the following requirements: a. White blood cell count ≥3×109/L; b. Neutrophil count ≥1×109/L (no colony-stimulating factor treatment within 2 weeks prior to the examination); c. Hemoglobin ≥60g/L;
  2. Liver function: ALT≤3×ULN (except for elevated ALT caused by inflammatory myopathy); AST≤3×ULN (except for AST elevation caused by inflammatory myopathy); TBIL≤1.5×ULN (except for Gilbert's disease).

     TBIL≤1.5×ULN (except Gilbert's syndrome, total bilirubin≤3.0×ULN);
  3. Renal function: creatinine clearance (CrCl) ≥ 30 ml/minute (Cockcroft/Gault formula, except for disease-induced decline in CrCl);
  4. Coagulation: international normalized ratio (INR) ≤ 1.5 x ULN, prothrombin time (PT) ≤ 1.5 x ULN.
  5. Cardiac function: hemodynamic stability;
* female subjects of childbearing potential and male subjects with a partner of childbearing potential are required to use medically approved contraception or be abstinent from sexual intercourse for at least 6 months during and after study treatment; female subjects of childbearing potential must have had a negative serum HCG test within 7 days prior to study enrollment and must not be breastfeeding;
* Voluntarily participate in this clinical study and sign the informed consent form, good compliance and cooperate with follow-up visits.
* Specific inclusion criteria:
* Relapsed refractory systemic lupus erythematosus.
* meets the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE;
* have a Disease Activity Score SLEDAI⁃2000 ≥ 6; and have at least one British Isles Lupus Assessment Group Index (BILAG-2004) Category A (severe manifestations) or two Category B (moderate manifestations) organ scores, or both; or have a Disease Activity Score SLEDAI-2000 ≥ 8;
* Definition of relapse-refractory: failure of conventional treatment for more than 6 months or recurrence of disease activity after remission.
* Relapsing Refractory/Progressive Diffuse Systemic Sclerosis
* meets the 2013 ACR's classification criteria for systemic sclerosis consistent with a diffuse presentation
* is positive for antibodies related to systemic sclerosis;
* diffuse cutaneous sclerosis manifestations or active interstitial lung disease (HRCT suggestive of ground-glass exudates);
* definition of relapsing-refractory: failure of conventional treatment for more than 6 months or recurrence of disease activity after remission.
* Definition of Progressive: Rapid cutaneous progression (>25% increase in mRSS); or pulmonary progression (10% decrease in FVC, or >5% decrease in FVC with 15% decrease in DLCO).
* Note: It is sufficient if one of Articles 4 and 5 is fulfilled.
* Relapsed refractory/progressive inflammatory myopathy
* meets the 2017 EULAR/ACR classification criteria for inflammatory myopathies (including DM , PM, ASS, and NM);
* is positive for antibodies to myositis;
* in those with muscle involvement, an MMT-8 score of less than 142 and abnormal findings on at least two of the following five core measurements (PhGA, PtGA, or Extramuscular Disease Activity Score ≥2; Total HAQ Score ≥0.25); Myosin level 1.5 times the upper limit of the normal range); or MMT-8 ≥142 in the presence of active interstitial lung disease (HRCT suggestive of ground-glass exudates);
* Definition of relapse refractory: failure of conventional treatment for more than 6 months or recurrence of disease activity after remission.
* Definition of progressive: the presence of exacerbation of myositis or rapidly progressive interstitial pneumonia.
* Note: It is sufficient if one of Articles 4 and 5 is fulfilled.
* Relapsed Refractory/Progressive Immune Thrombocytopenia
* meets the 2019 American Society of Hematology (ASH) classification criteria for immune thrombocytopenia;
* have bone marrow morphology characterized by increased or normal megakaryocytes with impaired maturation;
* exclude other secondary thrombocytopenia
* Definition of recurrent refractory: a patient who fails to achieve a satisfactory outcome after first-line standard therapy (e.g., glucocorticoids), including a full dose and course of therapy, i.e., platelet counts that cannot be maintained at a safe level (generally considered to be platelet counts > 30 × 10⁹ /L and without overt bleeding symptoms).
* Definition of progressive: a sustained decline in platelet count over the course of the disease, or a progressive worsening of bleeding symptoms, which may be accompanied by signs such as splenomegaly, and a progressively worse response to conventional therapy.
* Note: It is sufficient if one of Articles 4 and 5 is fulfilled.

Exclusion Criteria:

* A history of severe drug allergies or sensitivities;
* the presence or suspicion of fungal, bacterial, viral or other infections that are uncontrolled or require treatment
* persons with central nervous system disorders caused by ADs or not caused by ADs.
* those with intolerable cardiac function;
* subjects with congenital immunoglobulin defects.
* history of malignant tumors within the last five years.
* end-stage renal failure;
* subjects with positive Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA titer higher than the upper limit of the test; subjects with positive antibody to Hepatitis C virus (HCV) and peripheral blood HCV RNA; subjects with positive antibody to Human Immunodeficiency Virus (HIV); and subjects with a positive test for Syphilis;
* mental illness and severe cognitive impairment;
* have participated in other clinical trials within 3 months prior to enrollment;
* immunosuppressants or biologics with a therapeutic effect for the indication within five half-lives prior to enrollment
* women who are pregnant or intend to become pregnant;
* subjects who, in the opinion of the investigator, have other reasons for not being included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
chimeric status | 1 year after transplantation
  Detecting the chimerism in recipients' peripheral blood and bone marrow.Chimerism is generally measured in percentages(%)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 155, The First Affiliated Hospital of China Medical University, Nanjing North Street, Heping District, Shenyang, Liaoning Province, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Share IPD with The First Affiliated Hospital of China Medical University
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study will run from August 2025 to August 2027.
Access Criteria: The sponsors and collaborators are able to access the IPD and supporting information, IPD relies on team collaboration , as well as continuous improvement in innovation and efficiency. Participants will share project information, including the project's objectives, statistical datas, and clinical study report.